CLINICAL TRIAL: NCT01363934
Title: A Dose-Block Randomized, Double-blind Placebo Controlled, Open-label Active Controlled, Dose-escalation Study to Investigate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of GC1113 After Single Intravenous/Subcutaneous Administration in Healthy Male Subjects
Brief Title: To Evaluate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of Erythropoietin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Collaborators: Symyoo (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GC1113_P1
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Volunteer
Keywords: Erythropoietin; EPO-hFC
MeSH Terms: interventions — GC1113; Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Group A (Experimental): GC1113 or Placebo: GC1113 0.3ug/kg to 5ug/kg once intravenously
  Interventions: Drug: GC1113
- Group B (Experimental): GC1113 or Placebo: GC1113 0.3ug/kg to 5ug/kg once intravenously
  Interventions: Drug: GC1113
- Group C (Experimental): GC1113 or Placebo: GC1113 0.3ug/kg to 5ug/kg once intravenously
  Interventions: Drug: GC1113
- Group D (Experimental): GC1113 or Placebo: GC1113 0.3ug/kg to 5ug/kg once intravenously
  Interventions: Drug: GC1113
- Darbepoetin alfa 30ug/kg by IV (Active Comparator): Darbepoetin alfa 30ug/kg once intravenously
  Interventions: Drug: Darbepoetin alfa
- Group H (Experimental): GC1113 or Placebo: GC1113 1ug/kg to 8ug/kg once subcutaneously
  Interventions: Drug: GC1113
- Group I (Experimental): GC1113 or Placebo: GC1113 1ug/kg to 8ug/kg once subcutaneously
  Interventions: Drug: GC1113
- Group J (Experimental): GC1113 or Placebo: GC1113 1ug/kg to 8ug/kg once subcutaneously
  Interventions: Drug: GC1113
- Group K (Experimental): GC1113 or Placebo: GC1113 1ug/kg to 8ug/kg once subcutaneously
  Interventions: Drug: GC1113
- Darbepoetin alfa 30ug/kg by SC (Active Comparator): Darbepoetin alfa 30ug/kg once subcutaneously
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: GC1113 — Each Group volunteers (n=10) will be administered GC1113 0.3ug/kg to 5ug/kg or Placebo (GC1113:placebo=8:2) once intravenously.
  Each Group volunteers (n=10) will be administered GC1113 1ug/kg to 8ug/kg or Placebo (GC1113:placebo=8:2) once subcutaneously.
  Arms: Group A; Group B; Group C; Group D; Group H; Group I; Group J; Group K
Drug: Darbepoetin alfa — Each Group volunteers (n=8) will be administered Darbepoetin alfa by IV or SC.
  Arms: Darbepoetin alfa 30ug/kg by IV; Darbepoetin alfa 30ug/kg by SC

SUMMARY:
This is a Dose-Block Randomized, Double-blind Placebo controlled, Open-label Active controlled, Dose-escalation Study to investigate the safety, tolerability, and Pharmacokinetics/Pharmacodynamics of GC1113 after Single Intravenous/Subcutaneous Administration in Healthy Male Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adult male subjects between 20 to 55 years of age
* 60kg ≤ weight ≤ 90kg, 19 ≤ BMI ≤ 27
* 12 g/dL ≤ Hemoglobin ≤ 16 g/dL within the 28 days prior to investigational product (IP)injection
* WBC ≥ 3.0Ⅹ10^9/L, platelet ≥ 140Ⅹ10^9/L within the 28 days prior to IP injection

Exclusion Criteria:

* Allergic to IP ingredients
* History of uncontrolled liver, kidney, respiratory, endocrine, neurology, immunology, hematology, mental symptom, circulatory and malignancy disease
* Prior exposure to EPO, darbepoetin, other EPO, immunoglobulin, IV iron supplementation
* History of hypersensitivity reaction to EPO, darbepoetin, excipient of IP or hyperergia to iron supplementation
* Epilepsy within the 6 months prior to IP injection
* Positivity for HIV antibody, HBsAg, HCV antibody test
* Spleen length > 16㎝

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety/ Tolerability Evaluation | Up to 29 days after investigational product administration
  Number of subjects with Adverse events, Physical examinations, Vital signs, electrocardiogram (ECG), Laboratory tests (including hematology, chemistry, coagulation, urinalysis)

SECONDARY OUTCOMES:
AUClast of GC1113, Cmax of GC1113 | Up to 29 days after investigational product administration
  Blood test, urinalysis, hemoglobin, reticulocyte count, reticulocyte hemoglobin contents
Immunogenicity of GC1113 | Up to 29 days after investigational product administration
  Antibody (GC1113) test
To compare safety and Pharmacokinetics/Pharmacodynamics with active control | Up to 29 days after investigational product administration
  Abdominal Ultrasonograpy, egio genus radiology, blood test, urinalysis, hemoglobin, reticulocyte count, reticulocyte hemoglobin contents

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD., Ph.D, Principal Investigator — Seoul National University Hospital